CLINICAL TRIAL: NCT07378865
Title: A Phase 1, Open-label, Single-dose Study Evaluating the Excretion of Suzetrigine Into Breast Milk in Healthy Lactating Female Subjects
Brief Title: Evaluation of the Excretion of Suzetrigine Into Breast Milk in Healthy Lactating Female Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX25-548-021
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SUZ (Experimental): Participants will receive a single dose of SUZ on Day 1.
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Tablets for Oral Administration.
  Other Names: VX-548; SUZ; JOURNAVX

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK) of suzetrigine (SUZ) and its active metabolite in breast milk of lactating female participants. In addition, the purpose is also to evaluate the relative infant dose (RID), safety and tolerability of SUZ and its active metabolite in lactating female participants.

DETAILED DESCRIPTION:
The study is being conducted to evaluate the PK, safety and tolerability of SUZ and its active metabolite in lactating female participants.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index of greater than or equal to (≥) 18.0 to less than (<) 40.0 kilogram per meter square (Kg/m^2) at the Screening Visit
* Participants between 6 weeks and 12 months (inclusive) postpartum from a pregnancy of at least 37 weeks gestation, as of Day 1
* Willing to perform regular pumping to maintain milk supply for the duration of the study
* Participants with well-established lactation, defined as breastfeeding and/or pumping at least 3 times per day

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before study drug dosing
* History of breast implants, breast augmentation, or breast reduction surgery that significantly impacts breastfeeding or collection of milk from one or both breasts
* History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant
* Pregnant or planning to become pregnant during the study or within 30 days after receiving study drug

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Total Amount of SUZ in Breast Milk of Lactating Female Participants | From Day 1 up to Day 10
Total Amount of SUZ Metabolite in Breast Milk of Lactating Female Participants | From Day 1 up to Day 10
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of SUZ and its Metabolite in Breast Milk | From Day 1 up to Day 10
Maximum Observed Concentration (Cmax) of SUZ and its Metabolite in Breast Milk | From Day 1 up to Day 10

SECONDARY OUTCOMES:
RID of SUZ and its Metabolite From Breast Milk | From Day 1 up to Day 10
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 16

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/